CLINICAL TRIAL: NCT00006336
Title: Sensory Training for Treatment of Focal Dystonia
Brief Title: Sensory Training to Treat Focal Dystonia
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000227; 00-N-0227
Record Dates: First submitted 2000-10-04; First posted 2000-10-05 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2001-11

CONDITIONS: Dystonic Disorder
Keywords: Gap Detection Test; Fahn-Scale; Visual Analog and Verbal Scale; Writing Standard Paragraph; Braille Reading Grade I
MeSH Terms: conditions — Dystonic Disorders

SUMMARY:
This study will examine the effectiveness of Braille reading as a sensory training program for improving symptoms of focal (localized) dystonia, a movement disorder caused by sustained muscle contractions. Musicians, writers, typists, athletes and others whose work involves frequent repetitive movements may develop focal dystonia of the hand. Dystonia patients have an impaired sense of touch, and it is thought that symptoms may improve with sensory tactile (touch) training.

Patients with task-specific dystonia and healthy normal volunteers may be eligible for this 8-week study. Patients will undergo evaluation of their dystonia and a complete neurologic examination. Healthy volunteers will have a complete physical examination.

On the first day of the study, after 4 weeks and after 8 weeks, all participants will have a gap detection test for sensory perception testing. The test uses eight plastic devices called JVP-Domes with ridges of different widths on the surface. The subject's arm and hand are held in palm-up position and the right index finger is tested for about 1 second 20 times with each dome. The subject is asked to report whether the direction of the dome is vertical or horizontal. The test takes about 30 minutes. Patients with dystonia will also have a their symptoms evaluated at these visits. The evaluation involves completing a written questionnaire and writing a paragraph.

All participants will be trained in Braille reading at NIH. Sessions will be given every day the first week, twice a week the second and third weeks, and once a week the following weeks.

DETAILED DESCRIPTION:
It has been hypothesized that dystonia may be a sensory disorder. Animal studies as well as physiological studies of patients with focal dystonia have demonstrated sensory dysfunction. It has also been shown that patients with dystonia have impaired sensory perception including when assessed with the JVP gap detection test. This could possibly result from enlargement and dedifferentiation of representations in the sensory cortex. We therefore hypothesize that sensory training could improve the impaired sensory perception and hence improve the dystonia. This study will examine if Braille reading as a sensory training program can correct the sensory perception and the dystonia. The primary outcome is improvement in the JVP gap detection test.

ELIGIBILITY:
Patients with idiopathic task specific dystonia and healthy normal volunteers.

Patients must not be receiving botulinum-toxin treatment or other medications for the past three months prior to entering the study.

Patients must be able to keep their hand in a pronated 'reading' position for one hour.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22
Dates: Start 2000-09; Study Completion 2001-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Byl N, Wilson F, Merzenich M, Melnick M, Scott P, Oakes A, McKenzie A. Sensory dysfunction associated with repetitive strain injuries of tendinitis and focal hand dystonia: a comparative study. J Orthop Sports Phys Ther. 1996 Apr;23(4):234-44. doi: 10.2519/jospt.1996.23.4.234. PMID 8775368
- [Background] Bara-Jimenez W, Shelton P, Sanger TD, Hallett M. Sensory discrimination capabilities in patients with focal hand dystonia. Ann Neurol. 2000 Mar;47(3):377-80. PMID 10716260
- [Background] Bara-Jimenez W, Catalan MJ, Hallett M, Gerloff C. Abnormal somatosensory homunculus in dystonia of the hand. Ann Neurol. 1998 Nov;44(5):828-31. doi: 10.1002/ana.410440520. PMID 9818942